CLINICAL TRIAL: NCT03770156
Title: Attentats - Continuité Des Soins
Brief Title: Terrorist Attack - Continuity of Care
Acronym: CUMP75
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI18012J; 2017-A01382-51 (Other: ID-RCB)
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Stress Disorder; Major Depressive Episode
Keywords: Terrorist attack; Post-Traumatic Stress Disorder; Depression; Psychotherapy; Mental health; Victimology; Mourning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Psychological Well-Being | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects who contacted CUMP by phone: Subjects who contacted CUMP (Medical Psychological Emergency Cell) by phone from Paris November 13th, 2015, London 11th,2017 ; Barcelone 17-18th, 2017 ; Strasbourg 11th, 2018.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Overall Impression of the current state and evolution since the attacks

SUMMARY:
On November 13th 2015, a terrorist attack killed 129 victims in Paris. An emergency crisis unit (CUMP) has been activated in Paris in the days following the attack and a subunit was in charge to answer to the phone calls of victims and their relatives. The same emergency crisis unit have been activated for the terrorist attack in London, 2017 june 3, terrorist attack in Barcelone 2017 august 17-18, terrorist attack in Strasbourg 2018 December 11 The purpose of this observational study is to document the evolution of psychiatric symptoms among subjects who called the CUMP and to collect information about the type of medical or non-medical care they were seeking for.

DETAILED DESCRIPTION:
The care of the victims of natural disasters or mass disasters such as terrorist attacks is now better structured and organized. The efficacy of debriefing or of defusing has been and is still debated, sometimes bitterly. The aim of the present study is not to demonstrate utility or futility of such approaches, but to i) evaluate their global improvement over the past three years. ii) to list the type of support that the victims were seeking in their attempt to get rid of the symptoms which appeared after the terrorist attack of November 2015 in Paris.

iii) to collect their opinions about the way the CUMP (emergency medico-psychological unit of Paris, France) managed the support to the victims.

Participating subjects registered on the occasion of their first contact with the CUMP 75 by phone during the week following the attack

ELIGIBILITY:
Inclusion Criteria:

- All subjects who called the CUMP of Paris between November 13th, 2015 and January 31st, 2016; London 11th,2017 ; Barcelone 17-18th, 2017 ; Strasbourg 11th, 2018 and completed the questionnaire.

Exclusion Criteria:

- Subjects who did not consent to their participation to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who called the CUMP of Paris, London, Barcelone and Strasbourg after terrorist attacks were either direct, undirect victims or their relatives.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression - Improvement scale (CGI-I) | One day
  Self-assessment of improvement or aggravation

SECONDARY OUTCOMES:
Clinical Global Impression - Severity scale (CGI-S) | One day
  Self-assessment of symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Gaëlle ABGRALL-BARBRY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Gaëlle ABGRALL-BARBRY, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CUMP Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No